CLINICAL TRIAL: NCT02848976
Title: Re-training to Effort (RE) According to the Severity of Multiple Sclerosis: Preliminary Assessments Based on Fatigue and Quality of Life
Acronym: RE-SEP
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC13_0296
Record Dates: First submitted 2016-07-19; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- IA group: EDSS (Expanded Disability Status Scale) below 6 with RE
  Interventions: Other: Re-training to effort (RE)
- IB group: EDSS (Expanded Disability Status Scale) below 6 with no RE
- IIA group: EDSS (Expanded Disability Status Scale) betwin 6 and 8 with RE
  Interventions: Other: Re-training to effort (RE)
- IIB group: EDSS (Expanded Disability Status Scale) below 6 with RE
  Interventions: Other: Re-training to effort (RE)

INTERVENTIONS:
Other: Re-training to effort (RE) — The RE program includes three weekly sessions, supervised individually by a teacher in adapted physical activity, during 1:30, for four weeks, for a total of 12 sessions
  Groups: IA group; IIA group; IIB group

SUMMARY:
Regular physical activity promotes physical and mental well-being in the general population. Patients with multiple sclerosis (MS patients) tend them, to limit their physical activity or because of deficiencies related to the disease, or even on the advice of their caregivers in order to save their functional abilities. Time for leisure activity could be almost 20% lower in MS patients compared to healthy controls, and this situation is likely to aggravate the functional symptoms of multiple sclerosis.

The literature described the benefit of physical activity for MS patients according to protocols and varied assessments. Evaluations were indeed concern very analytical elements of metabolic functioning, nervous, muscular, cardiopulmonary etc ... or take into account the performance of components or fatigue and quality of life. Due to the multiplicity of RE protocols, sometimes on the verge of pragmatic goals of functional rehabilitation, the double issue was the profit earned by an RE program and of this benefit by level of severity of MS. The main objective of our study was an evaluation of the effects on fatigue and quality of life of a retraining program to effort suitable for levels of impairment and patients with MS activity limitations. The secondary objective was checking a performance improvement of the patients in this adapted program.

ELIGIBILITY:
Inclusion Criteria:

* Patients necessarily declare fatigue perceived as annoying in everyday life.
* Basic electrocardiogram should be absolutely normal.
* Patients should subject themselves to regular participation in the RE program

Exclusion Criteria:

* In the previous month the inclusion or during the RE, the MS patients should not have presented thrust nor undergone intravenous chemotherapy, or have been in care center.
* Free of cognitive impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Due to the double question about the expected benefits of our CR program, the inclusion of patients was conducted in two distinct periods, from specialized MS consultations in the services of Neurology and Physical Medicine and Rehabilitation ( MPR) of the University Hospital of Nantes (France). The first period (I) would lead to compare patients with EDSS less than 6 performing an exercise training (retrained group = IA) and patients with similar levels of EDSS not engaged in physical training (not retrained group = IB). The second period (II) compared to patients EDSS between 6 and 8 (EDSS group high = IIA) and patients with lower EDSS (EDSS group IIB = low), the two groups were following a RE program.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
SEP-59 questionnaire in MS | 1 month
  The first main criteria was established by the link between the quality of life (SEP-59 self-questionnaire scores) and the specific numerical data of multiple sclerosis
Scale impact of fatigue in MS (EMIF-SEP) | 1 month
  The second main criteria was established by the link between the fatigue (scale impact of fatigue in MS (EMIF-SEP), self-questionnaire scores) and the specific numerical data of multiple sclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Marc LE FORT, Doctor, Principal Investigator — Nantes University Hospital
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No